CLINICAL TRIAL: NCT07395284
Title: The Effect of Gamified Metaverse-Based Training on Nursing Students' Self-Efficacy and Metaverse Perception Regarding Pressure Injury Management: A Randomized Controlled Study
Brief Title: The Effect of Gamified Metaverse-Based Training on Nursing Students' Self-Efficacy and Metaverse Perception Regarding Pressure Injury Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, BETUL SAHIN KILINC, lecturer, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17162298.600-373
Record Dates: First submitted 2026-01-21; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Pressure Ulcers, Bedsores, Decubitus Ulcer; Nursing Education; Gamification; Self-Efficacy
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified metaverse-based educational application (Experimental): Gamified metaverse-based educational application
  Interventions: Behavioral: Gamified metaverse-based educational application
- Traditional-based education practice (No Intervention): traditional-based education practice

INTERVENTIONS:
Behavioral: Gamified metaverse-based educational application — Students in the intervention group will receive gamified metaverse-based training.
  Arms: Gamified metaverse-based educational application

SUMMARY:
Introduction: Pressure ulcers are a largely preventable clinical problem that negatively impacts the quality of patient care and constitutes a significant economic burden for healthcare systems. The prevention and effective management of these ulcers are closely related to nurses' knowledge, skills, and self-efficacy levels. However, current nursing education programs show a limited number of practice-based and interactive training approaches for the prevention and management of pressure ulcers. In recent years, innovative and technology-supported training methods such as gamification and metaverse have emerged as promising approaches for improving students' knowledge and self-efficacy levels by increasing their active participation in learning processes. Aim: The aim of this research is to evaluate the effect of gamified metaverse-based training developed for nursing students on their knowledge level, academic self-efficacy, and metaverse perception regarding pressure ulcer management.

Method: The research was planned as a randomized controlled experimental design. The population of the study will consist of students studying in the nursing department. The sample size was calculated using G*Power based on PUKAT 2.0-T scores; Assuming a two-way α=0.05 and power=0.80, at least 26 participants were selected for each group, and the total sample size was planned as 60 students, taking into account possible losses. Participants will be administered a Demographic Information Form, the Pressure Ulcer Knowledge Level Assessment Tool 2.0-Updated Version (PUKAT 2.0-T), and the Nursing Students Academic Self-Efficacy Scale. Participants will be randomly assigned to intervention and control groups based on their pre-test scores. The intervention group will receive traditional classroom theoretical training and gamified metaverse-based training for two weeks, while the control group will receive traditional classroom theoretical training. Post-tests will be administered immediately after the intervention and one month later. In addition, the Metaverse Perception Scale will be administered to the intervention group. Data will be collected using the Pressure Ulcer Knowledge Assessment Tool 2.0-Updated Version (PUKAT 2.0-T), the Nursing Students Academic Self-Efficacy Scale, and the Metaverse Perception Scale for Nursing Students.

Results: The obtained data will be analyzed using appropriate statistical methods.

Conclusion: This research is expected to provide evidence regarding the effectiveness of innovative digital education models in nursing education and contribute to the development of educational strategies for the prevention of pressure ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate in the research,
* Be a second-year undergraduate nursing student,
* Be able to understand and speak Turkish,
* Have healthy hearing, vision, and speech.

Exclusion Criteria:

* The student voluntarily requesting to withdraw from the study
* The student ceasing to use the metaverse domain during the study period
* Completing the survey form incompletely.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Pressure Ulcer Knowledge Assessment Tool 2.0 - Updated Version (PUKAT 2.0-T) | Before the intervention, within 1 hour after the intervention, and one month after the intervention.
  PUKAT 2.0 is a multiple-choice, true-false scored measurement tool. This test was developed by Manderlier et al. (2017) to determine nurses' knowledge level regarding pressure ulcers and adapted into Turkish by Dalli et al. (2022). The test addresses knowledge level regarding pressure ulcers within six themes and contains a total of 25 questions. The score ranges from 0 to 25. According to the validity and reliability study results of the Turkish version of the test; (1) content validity index is 0.90, (2) test-retest reliability is 0.83 (between 0.70-0.92 for sub-themes), (3) item difficulty indices range from 35-75%, (4) item discrimination indices range from 0.44-0.92, and (5) internal consistency (Cronbach's alpha) value is 0.72. Necessary permissions for the use of the measurement tool have been obtained from its developers.
Academic Nurse Self-Efficacy Scale | Before the intervention, within 1 hour after the intervention, and one month after the intervention.
  The scale developed by Bulfone et al. (2019) to determine the academic self-efficacy of undergraduate nursing students consists of 14 items and four sub-dimensions. The scale comprises the following sub-dimensions: internal emotion management (items 1, 2, 3), self-control behavior (items 4, 5, 6, 7), external emotion management (items 8, 9, 10, 11), and sociability (items 12, 13, 14). The items on this scale are scored between 1 and 5, and the question "How confident are you?" is scored using a 5-point Likert scale (1 = I have no confidence in myself, 5 = I have a lot of confidence in myself). As the scores obtained from the scale increase, the academic self-efficacy of nursing students increases. There are no items in the scale that are reverse-scored. The Cronbach alpha value of the original scale is 0.84, while in this study it is 0.82.

SECONDARY OUTCOMES:
Metaverse Perception Scale for Nursing Students | within 30 minutes after intervention
  To evaluate the metaverse perception levels of nursing students, the Metaverse Perception Scale for Nursing Students, developed by Yıldırım and Karaman (2024), will be used. The scale consists of a total of 24 items and includes four sub-dimensions: Education (items 1-9), Technology (items 10-14), Challenges (items 15-19), and Lifestyle (items 20-24). The scale items will be rated on a 5-point Likert scale, with response options ranging from "1=Strongly Disagree" to "5=Strongly Agree". A high score obtained from the scale will indicate a high metaverse perception. Items belonging to the Challenges sub-dimension will be reverse-coded to calculate the average score, while the average score for the entire scale will be evaluated without reverse coding. The overall reliability coefficient of the scale is reported to be Cronbach's alpha=0.955, while the Cronbach's alpha values for the sub-dimensions range from 0.930 to 0.955.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Ankara, Turkey (Türkiye)